CLINICAL TRIAL: NCT07008612
Title: Characterisation of Language and Prosody Disorders, Cognitive Functioning and Behavioural Problems in MYT1L Syndrome
Brief Title: MYT1L Syndrome: a Rare Paediatric Genetic Syndrome Responsible for a Neurodevelopmental Disorder
Acronym: MYT1L
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/0255/OB; IDRCB : 2024-A02492-45 (Other: ANSM)
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: MYT1L Syndrome
Keywords: combination of symptoms and physical features which are found together in a person and are all due to the same underlying cause

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Patients with a genetic syndrome linked to the MYT1L gene — * Neuropsychological assessment by the neuropsychologist (lasting 1h30)
  * Speech and language assessment (including language and prosody) by the speech therapist, lasting 1h30
Diagnostic Test: Patients with a neurodevelopmental disorder of genetic origin but not linked to MYT1L — Evaluation de la prosodie par l'orthophoniste (45 minutes)

SUMMARY:
MYT1L syndrome is a rare genetic syndrome, recently described in 2011, with paediatric onset, responsible for a neurodevelopmental disorder combining psychomotor retardation, learning difficulties and/or intellectual development disorders, epilepsy, overweight and eating disorders. The Rouen genetics department is currently positioned as a clinical expert in this disease.

The study published in 2020 by our team (Coursimault J et al., Hum Genet. 2022, PMID: 34748075) has enabled us to describe 40 new individuals worldwide, to gain a better understanding of this disease, to specify the genotype-phenotype relationships and to describe new clinical signs. We were able to confirm the presence of a neurodevelopmental disorder in 100% of patients, which includes: language delay, impaired orality, global and facial hypotonia, prosodic features and behavioural problems. This will be the first study in the world to characterise the neuropsychological, language and prosodic profiles of MYT1L patients.

DETAILED DESCRIPTION:
Although neuropsychological and speech therapy assessment is part of the routine work-up of any patient with a neurodevelopmental disorder, the heterogeneous use of assessment scales has not made it possible to obtain a precise characterisation of the neuropsychological and language profile of patients with MYT1L syndrome in retrospective studies. As a result, it is not possible to establish specific language and behavioural rehabilitation treatments. The aim of the study is to provide substantiated information on language (oral language, speech), prosody (reception and expression) and cognitive-behavioural aspects (global IQ, executive functions, sensory profile, attention, aggression, intolerance to frustration, anxiety). This project proposes to carry out a protocol used in routine care to assess language, prosody, cognitive functions and mood disorders, with the aim of identifying a specific language, prosody, cognitive and behavioural profile of patients with MYT1L syndrome, which could lead to better assessment in the future, screening for disorders and better targeting of rehabilitation in future patients, and to identify profiles suggestive of MYT1L syndrome in patients who have not had genetic confirmation (no variation identified or variation of uncertain significance).

ELIGIBILITY:
Inclusion Criteria:

MYT1L Group Patients

* Minimum age for inclusion: 6 years
* Maximum age for inclusion: no upper age limit
* Language: French
* Consent of parents or legal guardian
* Social security coverage required

Prosody Group Patients

* Unaided visual or hearing impairment making assessments impossible
* Non-French speaking patients
* Patients with a dual molecular genetic diagnosis also causing a neurodevelopmental disorder
* Acquired neurological disorder

Exclusion Criteria:

MYT1L Group patients

* Unaided visual or hearing impairment making assessments impossible
* Non-French speaking patients
* Patients with a dual molecular genetic diagnosis also causing a neurodevelopmental disorder
* Acquired neurological disorder

Prosody Group Patients

* Patients with molecularly confirmed MYT1L syndrome.
* Nonverbal patients

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult patients with MYT1L syndrome
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Speech-language profile | At enrollment visit
  Evaluation of the neuropsychological profile during an interview with the neuropsychologist allowing the administration of standardized tests completed with the patient and through questionnaires completed by the family

SECONDARY OUTCOMES:
Speech-language profile | At enrollment visit
  Assessment of the language profile through standardized tests completed with the patient during the interview with the speech therapist and questionnaires completed by the family
Prosodic speech therapy profile (patients with MYT1L syndrome) | At enrollment visit
  Evaluation of the prosodic profile of patients with MYT1L syndrome by voice recordings
Prosodic speech therapy profile (patients with a molecular diagnosis other than MYT1L) | At enrollment visit
  Evaluation of the prosodic profile of patients with a molecular diagnosis other than MYT1L by voice recordings

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: Yes
The data provided will be the property of the sponsor and will be used solely for its own research activities.